CLINICAL TRIAL: NCT06337656
Title: Influence of an Alternating Whole-Body Vibration Training on Muscle Mass and Muscle Strength in Patients With Liver Cirrhosis and Sarcopenia: A Clinical Pilot Project
Brief Title: Vibration Training Approach in Liver Cirrhosis
Acronym: VITAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Eva Dittmann, Principal Investigator, University Hospital of Cologne
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VITAL_0
Record Dates: First submitted 2024-03-03; First posted 2024-03-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Liver Cirrhosis
Keywords: Sarcopenia
MeSH Terms: conditions — Liver Cirrhosis; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Galileo Intervention (Experimental)
  Interventions: Device: Galileo WBV
- Galileo Control (No Intervention)

INTERVENTIONS:
Device: Galileo WBV — Side-Alternating Whole-Body Vibration Training
  Arms: Galileo Intervention

SUMMARY:
* Comprehensive Investigation of the Impact of Side-Alternating Whole-Body Vibration Training on Muscle Mass and Muscle Strength in Patients with Liver Cirrhosis and Sarcopenia
* Simultaneous Characterization and Evaluation of Dynamic Changes in Health-Related Quality of Life in our Patient Cohort with Liver Cirrhosis and Sarcopenia through Side-Alternating Whole-Body Vibration Training.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed or newly diagnosed compensated liver cirrhosis suffering from sarcopenia (combined decrease in muscle mass and muscle strength)
* The liver cirrhosis is in a compensated stage.
* The following etiologies of chronic liver disease are present: chronic hepatitis B infection, chronic hepatitis C infection, alcoholic liver disease, autoimmune hepatitis, cholestatic liver disease (PBC, PSC), or other chronic hepatopathy.
* Alcohol abstinence of at least 3 months in cases of alcohol-related liver disease.
* Routine cancer screening for the presence of a liver tumor (HCC surveillance) is routinely performed using MRI or CT scans, as ultrasound assessment is severely limited.
* Permission from the treating physician to engage in physical activity.
* Signed informed consent form.

Exclusion Criteria:

* Non-compliance with inclusion criteria
* Patients with recent hospitalizations (within the last 3 months) due to gastrointestinal bleeding, hepatic encephalopathy, or spontaneous bacterial peritonitis
* Presence of inadequately treated portal hypertension
* Known chronic liver disease not described in the above groups
* Alcohol consumption >20 g per day
* Excessive alcohol consumption during the study period leads to exclusion from the study
* Substance abuse
* Taking medications known to affect muscle mass or strength (e.g., Amiodarone, Chloroquine, Macrolides)
* Taking medications known to cause movement disorders (e.g., Reserpine, Lithium, Cyclosporine A, Dopamine agonists)
* Patients with unstable cardiovascular diseases: e.g., unstable angina pectoris, uncontrolled hypertension (≥ 160/100 mmHg), uncontrolled diabetes (blood sugar > 250 mg/dl), history of myocardial infarction or stroke
* Patients with musculoskeletal deformities, symptomatic rheumatoid or osteoarthritis
* Patients with untreated or newly diagnosed active malignant tumors in history
* Patients with neuromuscular or neurodegenerative diseases
* Patients with untreated hernias
* Patients with symptomatic, known untreated aortic aneurysm, with recent hospitalizations (within the last 6 months)
* Patients with fractures within the last 12 months
* Participation in moderate-intensity training programs for more than 2 hours per week
* Patients who have received chemotherapy at the time of the study or in the past 3 months
* Other underlying conditions that contraindicate vibration training and/or functional performance tests
* Circumstances preventing the individual from assessing the nature, scope, and possible consequences of the clinical trial
* Signs indicating that the subject is likely not to adhere to the study protocol (e.g., lack of cooperation)

  a. Definition of hepatic decompensation
* Occurrence of symptomatic ascites, hepatic encephalopathy, portal hypertensive bleeding (e.g., esophageal variceal bleeding), infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Effectiveness on muscle strength | 6 months
  Evaluation of the effectiveness of the intervention in terms of muscle strength using the hand-grip-strength
Evaluation of the Effectiveness on muscle strength | 6 months
  Evaluation of the effectiveness of the intervention in terms of muscle strength using the leg press
Evaluation of the Effectiveness on muscle strength | 6 months
  Evaluation of the effectiveness of the intervention in terms of muscle strength measuring the gait speed
Evaluation of the Effectiveness on muscle strength | 6 months
  Evaluation of the effectiveness of the intervention in terms of muscle strength measuring the Timed-Up-And-Go-Test
Evaluation of the Effectiveness on muscle mass | 6 months
  Evaluation of the Effectiveness on muscle mass through quantification of muscle mass by the skeletal muscle index (SMI) at the level of lumbar vertebral body 3 measured in MRI or CT.
Evaluation of the Effectiveness on muscle thickness | 6 months
  Evaluation of the Effectiveness on muscle mass through quantification of muscle mass by the transverse psoas muscle thickness (TPMT) at the level of lumbar vertebral body 3 measured in MRI or CT.
Evaluation of the Effectiveness on mobility, in particular the risk of falling | 6 months
  Evaluation of the Effectiveness on mobility, in particular the risk of falling by using the Tinetti test
Evaluation of the Effectiveness on physical function | 6 months
  Evaluation of the Effectiveness on physical function by using the Liver-Frailty-Index

SECONDARY OUTCOMES:
Evaluation of Safety of the Training Method | 12 weeks
  Evaluation of the safety of the training method by recording adverse events
Health-Related Quality of Life | 6 months
  Determination of Health-Related Quality of Life by using the Sarcopenia and Quality of Life (SarQoL®) questionnaire. The Sarcopenia and Quality of Life Questionnaire (SarQoL®), a specific questionnaire for assessing quality of life in sarcopenia, consists of 55 items, grouped into 22 questions rated on a 4-point Likert scale. The questionnaire can be scored up to 100 points, with a higher score reflecting a higher quality of life.
Health-Related Quality of Life | 6 months
  Determination of Health-Related Quality of Life by using the Short Form 36 (SF 36) questionnaire. The possible score ranges from 0 to 100 points, where 0 points represent the greatest possible health impairment, while 100 points indicate no health impairment.